CLINICAL TRIAL: NCT01398124
Title: A Pilot Study of Cyclin B1 Peptide-Pulsed Autologous Dendritic Cell Vaccine for Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: Cyclin B1 Peptide-Pulsed Autologous Dendritic Cell Vaccine for Resectable Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We will not be pursuing this study.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Chandra P. Belani, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-008
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: early stage non-small cell lung cancer; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Cyclin B1 Peptide — vaccine

SUMMARY:
Despite recent advances in the treatment of patients with resected NSCLC, disease recurrence and mortality related to lung cancer are common among patients with early stage non-small cell lung cancer (NSCLC). Therefore novel approaches are necessary to improve the outcome for early stage NSCLC. The preclinical studies conducted with vaccine based approaches provide the rationale to evaluate this as an adjunct to surgery for patients with early stage NSCLC. Administration of the vaccine before surgery will also allow for the evaluation of the tumor specimen for immunological responses to the vaccine.

DETAILED DESCRIPTION:
In the currently proposed study, patients will receive the first dose of the vaccine approximately 2 weeks prior to surgery. The second dose will be administered about 3-4 weeks following surgery. A booster dose of the vaccine will be given 6 months after the 2nd vaccine. The tumor tissue and serum will be studied for immunological responses following therapy with the vaccine. Patients are allowed to receive adjuvant chemotherapy if indicated. The choice of the chemotherapy regimen will be at the discretion of the treating physician, preferably 3-4 cycles of platinum combination regimen. The vaccine should be administered at least 2 weeks before chemotherapy is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer
* All patients must have one of the following stages: Stage IA(T1NO), and IB T2NO), II & IIIA (N2 negative)
* No prior chemotherapy or radiation therapy for non-small cell lung cancer
* Age >18 years
* ECOG performance status <2
* Patients must have acceptable organ and marrow
* Patient must be deemed surgically and medically resectable
* Men and women of childbearing potential must be willing to use effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients should not have received chemotherapy or radiotherapy within 3 months prior to entry to study.
* Patients with tumors involving the superior sulcus are not eligible.
* Patients must not have post-obstructive pneumonia or other serious infection at the time of registration or other serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Prior resection of lung cancer is allowed, if at least five years have elapsed between previous resection and registration.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Women of childbearing potential must have a negative pregnancy test.
* Known HIV-positive patients are excluded from the study.
* Patients with a history of known autoimmune disease are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ability of cyclin B1 peptide pulsed autologous dendritic cell vaccine to induce an immune response. | One week after second vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P. Belani, MD, Principal Investigator — Milton S. Hershey Medical Center